CLINICAL TRIAL: NCT00332124
Title: Double-blind Trial of Phosphatidylcholine During Pregnancy and Infant Serum Choline Levels
Brief Title: Safety and Effectiveness of Taking Choline Supplements During Pregnancy for Improving Infant Brain Development
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-0678; DATR A5-ETPD
Record Dates: First submitted 2006-05-30; First posted 2006-06-01 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Pregnancy; Child Development
MeSH Terms: interventions — Choline; lipostabil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Placebo Comparator): Participants will take placebo
  Interventions: Dietary Supplement: Placebo
- 2 (Active Comparator): Participants will take choline
  Interventions: Drug: Choline

INTERVENTIONS:
Drug: Choline — 900 mg every day until birth of infant
  Other Names: Polyenylphosphatidylcholine
  Arms: 2
Dietary Supplement: Placebo — Corn oil every day in place of choline
  Arms: 1

SUMMARY:
This study will evaluate the safety and effectiveness of taking choline supplements during pregnancy, and whether choline supplementation has an effect on infant development.

DETAILED DESCRIPTION:
Choline is an essential nutrient that can be found in foods, such as egg yolks, liver, and other meats. It is important for the composition and repair of normal cellular membranes, normal brain function, and normal cardiovascular function. Research has suggested that the presence of adequate amounts of choline during pregnancy and breastfeeding can help ensure healthy fetal brain development. Additionally, adequate prenatal choline levels may have long-lasting positive effects on cognitive function, including memory. However, sufficient research has not been done on the effects of choline on pregnant women and their unborn babies. This study will evaluate the safety and effectiveness of taking choline supplements during pregnancy, and whether taking choline during pregnancy will have an effect on infant development.

Participants in this double-blind study will be randomly assigned to receive either placebo or 900 mg of choline daily throughout pregnancy, until delivery. Babies will then begin receiving either placebo or choline daily from the time of birth until they are 3 months old. Participants will attend a baseline study visit that will include eligibility assessment, urine collection, measurement of vital signs, dispensing of study medication, and an ultrasound. Subsequent study visits will occur every 4 weeks throughout pregnancy and 6 months postpartum. Vital signs will be taken, urine samples will be collected, and study medication will be given at each visit. Two blood samples will be taken between Weeks 32 and 36 of gestation. Heel sticks will be performed on babies when they are 4 and 12 weeks old. Follow-up visits will be held every 6 months until the baby is 18 months old.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Between 10 and 18 weeks gestational age
* Healthy
* Diagnosis of psychosis

Exclusion Criteria:

* Use of any tobacco or nicotine product
* Drinks more than 1 alcoholic drink per day
* Use of illicit drugs
* History of trimethylaminuria
* History of kidney disease
* History of liver disease
* History of pre-pregnancy diabetes
* History of Parkinson's disease
* History of fetal death, fetal/infant congenital malformation, or fetal/infant genetic abnormality
* Evidence of noncompliance to study medication

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 351 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Sensory Gaiting (P50) | Measured at birth, 1 month and 3 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — University of Colorado, School of Medicine,
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Ross RG, Hunter SK, Hoffman MC, McCarthy L, Chambers BM, Law AJ, Leonard S, Zerbe GO, Freedman R. Perinatal Phosphatidylcholine Supplementation and Early Childhood Behavior Problems: Evidence for CHRNA7 Moderation. Am J Psychiatry. 2016 May 1;173(5):509-16. doi: 10.1176/appi.ajp.2015.15091188. Epub 2015 Dec 7. PMID 26651393
- [Derived] Ross RG, Hunter SK, McCarthy L, Beuler J, Hutchison AK, Wagner BD, Leonard S, Stevens KE, Freedman R. Perinatal choline effects on neonatal pathophysiology related to later schizophrenia risk. Am J Psychiatry. 2013 Mar;170(3):290-8. doi: 10.1176/appi.ajp.2012.12070940. PMID 23318559